CLINICAL TRIAL: NCT04095585
Title: Molecular Investigation, Using Chromosomal Microarray and Whole Exome Sequencing, of Patients Affected by Williams Beuren Syndrome and Autism Spectrum Disorder
Brief Title: Molecular Characterization of Patients Affected by Williams Syndrome and Autism.
Acronym: WBA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-WBA
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Williams Beuren Syndrome; Autism Spectrum Disorder
Keywords: Williams Beuren Syndrome; Autism Spectrum Disorder
MeSH Terms: conditions — Williams Syndrome; Autism Spectrum Disorder | interventions — Exome Sequencing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients presenting with WBS and ASD: patients with WBS and ASD. The diagnosis of WBS was confirmed by fluorescent in situ hybridization. All patients met formal ASD criteria.
  Interventions: Genetic: chromosomal microarray analysis (CMA) and whole exome sequencing (WES)

INTERVENTIONS:
Genetic: chromosomal microarray analysis (CMA) and whole exome sequencing (WES) — The investigator evaluated the following hypotheses:
  i) atypically large 7q11.23 deletions including additional genes; ii) rare pathogenic variants in genes located within the deletion, in particular GTF2I iii) additional pathogenic copy number variants (CNVs) or rare intragenic pathogenic variants located in other chromosomal regions with various inheritance patterns (autosomal recessive, X-linked, de novo autosomal dominant); given the small number of patients recruited, we focused on rare exonic variants considered to be pathogenic according to the criteria of the American College of Medical Genetics and Genomics (ACMG)

SUMMARY:
Williams Beuren syndrome (WBS) is a multiple malformations/intellectual disability (ID) syndrome caused by 7q11.23 microdeletion and clinically characterized by a typical neurocognitive profile including excessive talkativeness and social disinhibition, often defined as "overfriendliness" and "hypersociability". WBS is generally considered as the polar opposite phenotype to Autism Spectrum Disorder (ASD). Surprisingly, the prevalence of ASD has been reported to be significantly higher in WBS (12%) than in general population (1%). This study aims to investigate the molecular basis of the peculiar association of ASD and WBS. The investigator performed chromosomal microarray analysis and whole exome sequencing in six patients presenting with WBS and ASD, in order to evaluate the possible presence of chromosomal or gene variants considered as pathogenic.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of WBS was confirmed by fluorescent in situ hybridization.
* All patients met formal ASD criteria
* written informed consent

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with WBS and ASD.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Possible presence of pathogenic chromosomal | Day 0
  Assessed by chromosomal microarray analysis (CMA) and whole exome sequencing (WES) performed on DNA samples collected from the patients.
Possible presence of gene variants | Day 0
  Assessed by chromosomal microarray analysis (CMA) and whole exome sequencing (WES) performed on DNA samples collected from the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Rossi, MD, Principal Investigator — Hospices Civils de Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masson J, Demily C, Chatron N, Labalme A, Rollat-Farnier PA, Schluth-Bolard C, Gilbert-Dussardier B, Giuliano F, Touraine R, Tordjman S, Verloes A, Testa G, Sanlaville D, Edery P, Lesca G, Rossi M. Molecular investigation, using chromosomal microarray and whole exome sequencing, of six patients affected by Williams Beuren syndrome and Autism Spectrum Disorder. Orphanet J Rare Dis. 2019 May 31;14(1):121. doi: 10.1186/s13023-019-1094-5. PMID 31151468